CLINICAL TRIAL: NCT03362606
Title: Intervention of Ovarian Cancer Based on Engineered Immune Effectors (EIEs)
Brief Title: Engineered Immune Effectors Against Ovarian Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17018
Record Dates: First submitted 2017-11-20; First posted 2017-12-05 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Cytotoxic lymphocyte; OC-CTL
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OC-CTLs (Experimental): Autologous ovarian cancer specific cytotoxic lymphocytes
  Interventions: Biological: OC-CTLs

INTERVENTIONS:
Biological: OC-CTLs — 2 to 4 infusions, once a week, for 1x10^5~4x10^6 CTLs/kg via IV, abdominal cavity or tumor injection each time

SUMMARY:
This is a single-arm, open-label, phase I/II trial to evaluate the safety and efficacy of ovarian cancer specific cytotoxic lymphocytes (OC-CTLs) in women.

DETAILED DESCRIPTION:
Ovarian cancer is a cancer that forms in or on an ovary. The majority of ovarian cancers arise from the epithelium (outer lining) of the ovary. In 2015 it was reported found in 1.2 million women and resulted in 161,100 deaths worldwide. Among women it is the seventh-most common cancer and the eighth-most common cause of death from cancer. Treatment for ovarian cancer consists of surgery, chemotherapy, immunotherapy and sometimes, radiotherapy. The kind of treatment depends on many factors, including the type of ovarian cancer, its stage and grade, as well as the general health of the patient.

Adoptive immunotherapy with cytotoxic T lymphocytes (CTLs) reactive with specific viral antigens has proven to be effective. Here, the investigators aim to evaluate the safety and efficacy of multiple infusions of ovarian cancer specific cytotoxic T lymphocytes in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent obtained prior to any study-specific procedures.
2. Age older than 10 years.
3. Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1.
4. Expected survival ≥ 12 weeks.
5. Histologically confirmed and documented high risk International Federation of Gynecology and Obstetrics (FIGO): Stage II-IV.
6. Not pregnant, and on appropriate birth control if of childbearing potential.
7. Initial hematopoietic reconstitution with

   * neutrophils (ANC) ≥ 1,000/mm^3;
   * platelet (PLT) ≥ 100,000/mm^3.
8. Proper renal and hepatic functions (ULN denotes "upper limit of normal range") with

   * serum creatinine ≤ 2×ULN;
   * serum bilirubin ≤ 2×ULN;
   * AST/ALT ≤ 2×ULN;
   * ALKP ≤ 5×ULN;
   * serum bilirubin. 2.0 is acceptable in the setting of known Gilbert's syndrome.
9. Human immunodeficiency virus (HIV) and Hepatitis C virus (HCV) test were negative.

Exclusion Criteria:

1. Patients with ovarian tumors with low malignant potential (i.e. borderline tumors);
2. Patients with evidence of abdominal free air not explained by paracentesis or recent surgical procedure (prior, current or planned treatment).
3. Previous treatment of adoptive T cell therapy.
4. Current or recent treatment (within the 28-day period prior to Day 0) with another investigational drug
5. Minor surgical procedures within 2 days prior to Day 0 (including central venous access device placement for chemotherapy administration, tumor biopsies, needle aspirations).
6. Pregnant or lactating females.
7. Inadequate bone marrow function with

   * absolute neutrophil count < 1,000/mm^3;
   * platelet count < 100,000/mm^3;
   * Hb < 9 g/dL.
8. Inadequate liver and renal function with

   * serum (total) bilirubin > 1.5 x ULN;
   * AST & ALT > 2.5 x ULN (> 5 x ULN in patients with liver metastases);
   * alkaline phosphatase > 2.5 x ULN;
   * serum creatinine >2.0 mg/dl (> 177 μmol/L);
   * urine dipstick for protein uria should be < 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hour urine collection and must demonstrate < 1 g of protein/24 hr.
9. Serious active infection requiring i.v. antibiotics at during screening.
10. Subject infected with HCV (HCV antibody positive), HBV (HBsAg positive), and HIV (HIV antibody positive),Treponema pallidum antibody positive or TB culture positive.

Ages: 10 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Safety of OC-CTLs in patients using CTCAE version 4.0 standard to evaluate the level of adverse events | 6 months
  Physiological parameter (measuring cytokine response, fever, symptoms)

SECONDARY OUTCOMES:
Functional analyses of OC-CTLs in vitro | 4 weeks
  The specificity of OC-CTLs in vitro will be analysed by enzyme-linked immunospot assay (ELISPOT).
Anti-tumor effects | 1 year
  Objective response, such as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute; Qichun Cai, MD, Study Director — Jinshazhou Hospital of Guangzhou University of Chinese Medicine; Xun Lai, MD, Study Director — Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center
Locations (3):
- China (3):
  - Jinshazhou Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No